CLINICAL TRIAL: NCT01997437
Title: Clinical Trial Evaluation of Stem-cell Based Bioartificial Airway Transplantation for Patients With Benign and Malignant Laryngo-tracheal Diseases
Brief Title: Laryngo-Tracheal Tissue-Engineered Clinical Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuban State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11.G34.31.0065
Record Dates: First submitted 2013-11-05; First posted 2013-11-28 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-01

CONDITIONS: Tracheal Diseases
Keywords: Tissue-engineered tracheal transplantation
MeSH Terms: conditions — Tracheal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tissue-engineered airway transplantation (Other): Stem-cell seeded bioartificial tracheal scaffold
  Interventions: Device: Stem-cell seeded bioartificial tracheal scaffold

INTERVENTIONS:
Device: Stem-cell seeded bioartificial tracheal scaffold — Seeding the synthetic scaffold with autologous stem cells; scaffold' cultivation within 48-72 hours in bioreactor, injection of growth factors into scaffold in the first and last stages of the cultivation, replacement of the damaged trachea by generated tissue-engineered organ

SUMMARY:
The proposed protocol will involve the replacement of the trachea using a synthetic bioengineered scaffold seeded with autologous mononuclear cells as an intraoperative solution for patients with with benign and malignant laryngo-tracheal diseases or other terminal conditions of the trachea.

Tracheal transplant is indicated as the only therapeutic alternative in cases where instrumental, endoscopic and other evaluations show that the length of residual healthy airways (about 6 cm or longer than 50% of the airway length) and the localization and extension of the obstruction make it impossible to perform a surgical resection of the pathological segment.

In addition to tracheal surgical transplant techniques, this protocol requires knowledge and experience with autologous cell preparation as well as scaffold seeding procedures.

DETAILED DESCRIPTION:
Before transplantation the patients will have the laboratory and instrumental evaluations.

Three days before the transplantation the patient will be underwent bone marrow aspiration. The bone marrow mononuclear cells (MNC) will be isolated from the red blood cells (RBC) in the totally enclosed FDA approved automatic system (Sepax,BioSafe America, Inc.). The final product, re-suspended with cell culture medium (DMEM+10% albumin and 10% autologous plasma) in a volume of 200 mL, will be placed in a 600 mL transfer bag. 2 mL of the product will be taken from the bag before clinical use to test sterility using culture media and immunofluorescent cytometry to characterize cell type and viability.

Two days before the transplant, the patient will begin "boosting" therapy to mobilize cells by means of systemic injections of analogous recombinants of granulocyte colony-stimulating factor (GCSF)(Granocyte, 1 M IU/kg (max. 15 M IU) and Erythropoietin, 400 IU/kg (max.6,000IU). These will be injected for the two days prior to surgery.

InBreath Bioreactor (the special bioreactor for cultivating trachea) The work in the current protocol will involve a bioreactor design previously utilized by Macchiarini P. ang colleges in a successful first-in-man implantation of a tissue-engineered large airway replacement. The device, commercialized under the name, InBreath 3D Organ Bioreactor (Harvard Bioscience, Inc.) is designed for placement within a tissue culture incubator and consists of a modular polysulphone organ chamber, motor unit and remote controller. The chamber is easily detachable from the motor unit and its polysulphone construction permits sterilization with the standard gas plasma sterilization process that is readily available in the operating room in Peoria. The motor unit provides consistent rotation to the tissue holder within the chamber, ensuring controlled application of hydrodynamic shear forces to the developing tracheal construct. A fully enclosed motor housing protects the brushless motor from the corrosive moisture within the incubator. The remote control unit is placed outside the incubator providing a means to adjust rotational speed without disturbing the incubator environment.

The seeded construct was allowed to incubate in the bioreactor for 96 hours prior to removal for implantation. Based on the five previous adult cases using the POSS-PCU (Polyhedral oligomeric silsesquioxane-poly(carbonate-urea) urethane), PET(Polyethylene terephthalate) and PET:PU (Polyurethane) synthetic scaffolds, the internal and external surfaces of the scaffold will be seeded with the freshly isolated bone marrow mononuclear cell fraction. The bioreactor will be started with an initial speed of 0.5 cycles/min for 18 hours (then stepwise increase up to 2.5 cycles/min). Incubation will be during the 48 hours preceding the transplant procedure. This incubation protocol worked very well in the previous cases using the three different synthetic nanocomposite tracheal scaffolds.

Cultivation steps:

The tracheal reseeding procedure will be done in our aseptic culture GMP (Good Manufacturing Practice) facility that was established and fully functional.

1. Isolated MNC will be prepared according to the Sepax 2 protocol for bone marrow separation and resuspended in a 300ml bag containing 0.9%Normal saline solution (with 10% human albumin).
2. The sterilized scaffold (gamma irradiation sterilization), the bioreactor (plasma sterilization) and surgical instruments (autoclaved) will be placed into the laminar hood.
3. All persons that are manipulating the cells/bioreactor and scaffold will be fully trained in have GMP grade standards, namely sterile gloves, specific overalls, etc.
4. The bioreactor will be opened inside the hood in sterile conditions and placed on a sterile tissue. The scaffold will be mounted on the organ holding fixtures and placed into the bioreactor. Once the scaffold is transferred and fixed into the bioreactor the MNC (+DMEM plus albumin and autologous plasma) will be seeded on the scaffold´s surface. Medium (including autologous plasma and human albumin) will be added to the bioreactor chamber to a total volume of 200 ml.
5. The factors will add to medium: 39.3 ng/mL (100 nmol/L) dexamethasone, and 10 μg/mL insulin.
6. Then the bioreactor chamber (including the scaffold, MNC + 200 ml of medium) will be placed into the incubator and mounted onto the motor unit of the bioreactor (previously placed inside the incubator).
7. The bioreactor will be started with an initial speed of 0.5 cycle/min for 18h (then stepwise increase up to 2.5 cycles/min).
8. After 24h, an additional 50ml of the prementioned medium will be added to a total volume of 250ml inside the chamber. At this time a small aliquot of chamber fluid will be tested with gram stain and injected into culture media to check for contamination.
9. After 48 hours the chamber will be opened and an aliquot will harvested for culture and Gram stain. A small biopsy of the neotrachea will be taken for the MTT viability test. Once it is determined that the cells are viable and there is no sign of media contamination (Gram stain and interim reading of direct inoculation culture) the trachea will be deemed ready for implantation and the patient will be placed under anesthesia and the surgical procedure will be started.

Day of transplantation:

Intra-operative Surgical Procedure The morning of the transplant the graft will be tested for cell growth (MTT test and for sterility by gram stain and analysis of interim culture results). Once the graft is deemed ready for implantation, the patient will be placed under general endotracheal anesthesia.

Thoracic and abdominal procedures Having performed the resection of the airway's damaged segment, the airway construct will be seeded intraoperatively with the respiratory cell biopsies on the internal surface. The graft will be then injected (conditioned) with growth factors including 10 ng/mL of recombinant human transforming growth factor-β 3, 10 nmol/L recombinant parathyroid hormone-related peptide, 100 nmol/L dexamethasone, and 10 µg/mL insulin, GCSF (10 µg/kg) and Erythropoietin (40,000 UI) (to stimulate the mobilization of the peripheral hematopoietic cells). The implant will be then anastomosed proximally and distally so as to reconstruct the airway defect using sutures. It will be then covered and wrapped by an omentum major flap (adipose vascularized tissue detached from the large bend of the stomach, harvested on the right or left gastroepiploic artery and then carried over to the mediastinum trans-diaphragmatically or sub-sternally), to guarantee long-term protection of the graft and of the anastomosis and obtain indirect graft's neovascularisation.

After transplantation:

Post-operative treatment

To boost the regenerative process, the patient (current weight about 13 Kg) will be treated pharmacologically in the post-op period by systemic injections of:

1. Analogous recombinants of GCSF (Granocyte, 10 million IU/kg up to a maximum of 30 million IU)
2. Analogous synthetics of Erythropoietin (Epoetin alpha or beta 40,000 IU)

Both factors will be administered in suitable concentrations to stimulate the mobilization/recruitment of hematopoietic cells, in "regenerative" doses which have not been associated with any side-effects. Every second day the plasma Erythropoietin level and the blood count (including haemoglobin and white blood cell counts) will be monitored. Haemoglobin levels greater than 15 g/dl will raise concerns for hyper-viscosity and prompt removal of 10-20 cc/kg of blood and may prompt the addition of a continuous infusion of heparin to keep the Activated Partial Thromboplastin Time (APTT) levels between 40-60 seconds. White blood cell levels above 50-60,000/μl will be considered "toxic" and will result in a reduction/suspension of the GCSF therapy until numbers fall below 30,000. Treatment with GCSF and Erythropoietin will be carried out every other day for 2 weeks following the transplant according to the following table:

Follow-up

The follow-up will be carried out at the Cardiothoracic Surgery Department of the Krasnodar Regional Hospital, and will include:

1. Endoscopic evaluation (flexible and/or rigid bronchoscopy) of the transplanted airway every day for the first week and every other day for the second week, after which once a month for the first six months, and every 6 months thereafter for the first 5 years.
2. Evaluation of the blood count with white blood cell formula daily for the first two weeks.
3. Evaluation of mobilized progenitor cells from peripheral blood every second day during 2 weeks.
4. Immunogenic evaluation. After 3, 7 and 30 days from the transplant, a blood sample will be taken to make a study of the histocompatibility by evaluating the antibodies. The immunogenic follow-up will also be carried out after 3, 6 and 12 months from the transplant.
5. Post-operative Tobramycin inhalation (2x5ml/day for 30 days) to prevent from pneumonia and graft bacterial contamination.
6. Computerized tomography of the neck and chest with a three-dimensional reconstruction of the transplanted airway will be done at month 1, month 3 and month 6 of the follow-up, and every 6 months thereafter for the first 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Extended (> 60% total length) benign and malignant diseases
* Already maximally pretreated patients
* No absolute surgical contraindications
* No regional and/or micro-metastasis (BMB proven)
* Normal psychological or psychiatric habitus
* IRB, Ethics and National Transplant clearance
* Written informed consent

Exclusion Criteria:

* Presence of systemic metastatic lesions and positive mediastinal lymph nodes (malignancies);
* Routine functional and psychological contraindication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-12; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Macchiarini, MD, PhD, Principal Investigator — Kuban State Medical University
Locations (1):
- Clinical Regional Hospital #1, Krasnodar, Russia

REFERENCES:
- [Background] Jungebluth, P, Alici, E, Baiguera S, et al. Tracheobronchial transplantation with a stem-cell-seeded bioartificial nanocomposite: a proof-of-concept study. Lancet 2011 Dec 10; 378 (9808):1997-2004; Macchiarini P, Jungebluth P, Go T, et al. Clinical transplantation of a tissue-engineered airway. Lancet 2008; 372, 2023-3030; Acocella F, Brizzola S, et al. Prefabricated tracheal prosthesis with partial biodegradable materials: a surgical and tissue engineering evaluation in vivo. Journal of Biomaterials Science; Polymer Edition 2007; 18(5):579-594; Bader A, Macchiarini P. Moving towards in situ tracheal regeneration: the bionic tissue engineered transplantation approach. J Cell Mol Med 2010; 14(7):1877-89; Jungebluth P, Moll G, Baiguera S, Macchiarini P. Tissue engineered airway: a regenerative solution. Clin Pharm Ther 2012; 91:81-93;
- See also: Regeneration of airways and lung. The official website of the project "Investigating the molecular mechanisms and underlying pathways of regenerative medicine approaches the tissue-engineering and cell therapy of airways and lungs" — http://www.regmedgrant.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The dates of the recruitment period are from June 2012 to January 2014. The recruitment process have been done in medical clinic: Krasnodar Regional Hospital #1.
Groups:
- Stem-cell Seeded Bioartificial Trachea: Stem-cell seeded bioartificial tracheal scaffold: Seeding the synthetic scaffold with autologous stem cells; scaffold' cultivation within 48-72 hours in bioreactor, injection of growth factors into scaffold in the first and last stages of the cultivation, replacement of the damaged trachea by generated tissue-engineered organ
Period: Overall Study
Arm/Group | Stem-cell Seeded Bioartificial Trachea
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tissue-engineered Airway Transplantation
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 33 [28 to 41]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  Russian Federation | 5
  Jordan | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety of Stem-cell Seeded Bioartificial Tracheal Scaffold
Description: Safety of the tissue engineered trachea measured by occurrence of adverse events throughout 12 months post operative follow up
Time Frame: 12 months post operative follow up
Measure: Number; unit: participants
Arm/Group | Stem-cell Seeded Bioartificial Trachea
Number analyzed (Participants) | 6
participants | 0

2. Secondary Outcome: Number of Survival Patients
Description: To evaluate the survival of patient after transplantation of stem-cell seeded bioartificial trachea during 12 months post operative follow up.
Time Frame: 12 months post operative follow up
Measure: Number; unit: participants
Arm/Group | Stem-cell Seeded Bioartificial Trachea
Number analyzed (Participants) | 6
participants | 6

3. Secondary Outcome: Number of Disease Free Survival Patients
Description: The disease free survival of patient were evaluated after transplantation of stem-cell seeded bioartificial trachea during 12 months post operative follow up.
Time Frame: 12 months post operative follow up
Measure: Number; unit: participants
Arm/Group | Stem-cell Seeded Bioartificial Trachea
Number analyzed (Participants) | 6
participants | 6

4. Primary Outcome: Number of Mononuclear Cells (MNCs) Per ml
Description: MNCs were isolated from bone marrow fom each patient, and were counted by flow cytometry method. MNC were used for seeding on scaffold.
Time Frame: 1 time before seeding on scaffold
Measure: Mean (Standard Error); unit: MNCs per ml
Arm/Group | Stem-cell Seeded Bioartificial Trachea
Number analyzed (Participants) | 6
MNCs per ml | 2773000 (353579)

ADVERSE EVENTS:
Time Frame: 3 year
Description: Adverse events are assessed by physiological parameters, bronchoscopy with bronchoscopic alveolar lavage, computer tomography
Arm/Group | Stem-cell Seeded Bioartificial Trachea
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem-cell Seeded Bioartificial Trachea (N=6)
Granulation and Fistula (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Granulation or fistula resulted in 2 patient into re-transplantation, in 1 patient in explantation and tracheostoma

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No